CLINICAL TRIAL: NCT05828758
Title: Efficacy of Amoxicillin for Treatment of Enteral Nutrition Intolerance in Pediatric Intensive Care Unit
Brief Title: Amoxicillin for Enteral Nutrition Intolerance in Pediatric Intensive Care Unit
Acronym: AmoxENI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abanob Amgad Francis, Pediatric Resident, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Soh-Med-23-04-16MS
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Enteral Feeding Intolerance
Keywords: Feeding intolerance; Pediatric intensive care unit; PICU; Amoxicillin
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Two groups of children with enteral feeding intolerance:
  Study group: will receive amoxicillin 10 mg/kg (50 mg/ml concentration) by nasogastric tube 3 times daily (8 hours apart) 10 minutes before bolus gastric feeding for 7 days. The nasogastric tube will be flushed by 5 ml distilled water after each dose.
  Control group: will receive equal volume of distilled water (0.2 ml/kg + 5 ml) as a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Enrolled children will be equally randomized into study and control group using computer generated numbers, which will be sealed into sequentially numbered opaque envelopes by a person not belonging to the research team. For each enrolled participant, the envelope in order will be opened, and the assigned study drug will be used. A pharmacist will fill the active and placebo preparations in similar containers with sealed code for identification. Participants' families, treating clinicians, and investigators will be unaware of group assignment and drug/placebo therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children receiving amoxicillin
  Interventions: Drug: Amoxicillin
- Comparison group (Placebo Comparator): Children receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin 10 mg/kg (50 mg/ml concentration) by nasogastric tube 3 times daily (8 hours apart) 10 minutes before bolus gastric feeding for 7 days.
  Arms: Study group
Other: Placebo — Distilled water 0.2 ml/kg by nasogastric tube 3 times daily (8 hours apart) 10 minutes before bolus gastric feeding for 7 days.
  Arms: Comparison group

SUMMARY:
The goal of this randomized controlled study is to investigate the efficacy of enteral amoxicillin for the treatment of children with feeding intolerance in pediatric intensive care unit.

Children with feeding intolerance will be randomized into study and comparison groups. The study group will receive amoxicillin 10 mg/kg by nasogastric tube 3 times daily 10 minutes before bolus gastric feeding for 7 days. The comparison group will receive equal volume of distilled water as a placebo.

The primary outcome will be the improvement of feeding intolerance on day 7 study timepoint.

DETAILED DESCRIPTION:
Malnutrition is a common problem in critically ill children admitted to the pediatric intensive care unit (PICU) with a reported prevalence up to 57%. This condition is associated with increased length of hospital stay, morbidity (e.g., hospital-acquired infections, weakness, and longer duration of mechanical ventilation), and mortality. Data from observational studies indicate that adequate energy intake is associated with better outcomes in the PICU.

Enteral nutrition (EN) is the preferred route to administer nutritional support for critically ill children unless contraindicated. However, EN of critically ill children is challenging, and nutritional targets are commonly not attained.

EN intolerance (a clinical manifestation of delayed gastric emptying) is one of the main factors for limited delivery of enteral feeding. Promotility agents are commonly used as a first-line treatment for patients with EN intolerance. In critically ill adults, prokinetics have been shown to improve gastric emptying and enhance tolerance to gastric feeding. Available options include metoclopramide, domperidone, and erythromycin. However, there is insufficient evidence for recommending the use of prokinetics in children with critical illness to enhance gastric emptying and EN tolerance. Furthermore, currently available prokinetics are associated with serious side effects.

Amoxicillin/clavulanate combination is one of the most commonly prescribed antibiotics for children worldwide. Besides its antibacterial properties, some studies showed that amoxicillin/clavulanate could have prokinetic effects. However, well-designed randomized controlled trials to confirm the prokinetic effects of amoxicillin/clavulanate are lacking. Additionally, no human study has investigated the prokinetic effects of amoxicillin and clavulanate individually. In a study on juvenile rats, amoxicillin alone, but not clavulanate, was shown to increase the amplitude of spontaneous duodenal contractions. The use of amoxicillin alone rather than amoxicillin/clavulanate could have the advantages of avoiding the side effects of clavulanate, lowering the cost, and decreasing the risk of antibiotic resistance.

The goal of this randomized controlled study is to investigate the efficacy of enteral amoxicillin for the treatment of children with EN intolerance in PICU.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 1 month to 12 years.
* Nasogastric tube feeding
* Enteral nutrition intolerance after 7 days of admission to the PICU.

Exclusion Criteria:

* Failure to obtain informed consent.
* Allergy or contraindication to amoxicillin or other beta-lactam antibiotics.
* Current or recent (within 7 days) treatment with amoxicillin.
* Ongoing ketogenic diet.
* Clinical contraindications to advance EN feeds (e.g., bowel obstruction/tight stenosis, severe diarrhea/malabsorption, gut ischemia, severe hypoxemia/acidosis, intractable upper gastrointestinal bleeding, abdominal compartment syndrome, high-output fistula).

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Feeding tolerance on day 7 | 7 days
  Proportion of participants achieving feeding tolerance (enteral intake ≥ two-thirds of the prescribed daily target in the absence of gastrointestinal symptoms, including large gastric residual volume (≥ 50% of enteral feeding in the last 4 hours), vomiting (≥ 2 times gastric content in 24 hours period), diarrhea (≥ 4 times loose stool with negative fluid balance in 24 hours period), abdominal distention (≥ 2 cm increase in abdominal girth), abdominal pain, melena, or hematochezia) on day 7 study timepoint

SECONDARY OUTCOMES:
Enteral intake ≥ two-thirds of the prescribed daily target on day 7 | 7 days
  Proportion of participants achieving enteral intake ≥ two-thirds of the prescribed daily target on day 7 study timepoint
Change in achieved percentage of prescribed enteral feeding on day 7 study compared with baseline | 7 days
  Change in achieved percentage of prescribed enteral feeding on day 7 study timepoint compared with baseline
Large gastric residual volume on day 7 | 7 days
  Proportion of participants with large gastric residual volume (≥ 50% of enteral feeding in the last 4 hours) on day 7 study timepoint
Vomiting on day 7 | 7 days
  Proportion of participants with vomiting (≥ 2 times gastric content in 24 hours period) on day 7 study timepoint
Diarrhea | 7 days
  Proportion of participants with diarrhea (≥ 4 times loose stool with negative fluid balance in 24 hours period)
Abdominal distention | 7 days
  Proportion of participants with abdominal distention (≥ 2 cm increase in abdominal girth)
Melena/hematochezia | 7 days
  Proportion of participants with melena/hematochezia
Skin rash | 7 days
  Proportion of participants with skin rash

CONTACTS AND LOCATIONS:
Overall Officials: Safaa H Ali, MD, PhD, Study Chair — Sohag University
Locations (1):
- Pediatric Intensive Care Unit - Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data will be available after publication from the principal investigator upon a reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: After publication and for 3 years
Access Criteria: Through contacting the principal investigator by email

REFERENCES:
- [Background] Martinez EE, Douglas K, Nurko S, Mehta NM. Gastric Dysmotility in Critically Ill Children: Pathophysiology, Diagnosis, and Management. Pediatr Crit Care Med. 2015 Nov;16(9):828-36. doi: 10.1097/PCC.0000000000000493. PMID 26218259
- [Background] Eveleens RD, Hulst JM, de Koning BAE, van Brakel J, Rizopoulos D, Garcia Guerra G, Vanhorebeek I, Van den Berghe G, Joosten KFM, Verbruggen SCAT. Achieving enteral nutrition during the acute phase in critically ill children: Associations with patient characteristics and clinical outcome. Clin Nutr. 2021 Apr;40(4):1911-1919. doi: 10.1016/j.clnu.2020.09.005. Epub 2020 Sep 16. PMID 32981755
- [Background] Tume LN, Valla FV, Joosten K, Jotterand Chaparro C, Latten L, Marino LV, Macleod I, Moullet C, Pathan N, Rooze S, van Rosmalen J, Verbruggen SCAT. Nutritional support for children during critical illness: European Society of Pediatric and Neonatal Intensive Care (ESPNIC) metabolism, endocrine and nutrition section position statement and clinical recommendations. Intensive Care Med. 2020 Mar;46(3):411-425. doi: 10.1007/s00134-019-05922-5. Epub 2020 Feb 20. PMID 32077997
- [Background] Mehta NM, Skillman HE, Irving SY, Coss-Bu JA, Vermilyea S, Farrington EA, McKeever L, Hall AM, Goday PS, Braunschweig C. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Pediatric Critically Ill Patient: Society of Critical Care Medicine and American Society for Parenteral and Enteral Nutrition. Pediatr Crit Care Med. 2017 Jul;18(7):675-715. doi: 10.1097/PCC.0000000000001134. PMID 28691958
- [Background] Kratochvil M, Klucka J, Klabusayova E, Musilova T, Vafek V, Skrisovska T, Djakow J, Havrankova P, Osinova D, Stourac P. Nutrition in Pediatric Intensive Care: A Narrative Review. Children (Basel). 2022 Jul 11;9(7):1031. doi: 10.3390/children9071031. PMID 35884015
- [Background] Martinez EE, Pereira LM, Gura K, Stenquist N, Ariagno K, Nurko S, Mehta NM. Gastric Emptying in Critically Ill Children. JPEN J Parenter Enteral Nutr. 2017 Sep;41(7):1100-1109. doi: 10.1177/0148607116686330. Epub 2017 Jan 6. PMID 28061320
- [Background] Eveleens RD, Joosten KFM, de Koning BAE, Hulst JM, Verbruggen SCAT. Definitions, predictors and outcomes of feeding intolerance in critically ill children: A systematic review. Clin Nutr. 2020 Mar;39(3):685-693. doi: 10.1016/j.clnu.2019.03.026. Epub 2019 Mar 30. PMID 30962102
- [Background] Peng R, Li H, Yang L, Zeng L, Yi Q, Xu P, Pan X, Zhang L. The efficacy and safety of prokinetics in critically ill adults receiving gastric feeding tubes: A systematic review and meta-analysis. PLoS One. 2021 Jan 11;16(1):e0245317. doi: 10.1371/journal.pone.0245317. eCollection 2021. PMID 33428672
- [Background] Chiusolo F, Capriati T, Erba I, Bianchi R, Ciofi Degli Atti ML, Picardo S, Diamanti A. Management of Enteral Nutrition in the Pediatric Intensive Care Unit: Prokinetic Effects of Amoxicillin/Clavulanate in Real Life Conditions. Pediatr Gastroenterol Hepatol Nutr. 2020 Nov;23(6):521-530. doi: 10.5223/pghn.2020.23.6.521. Epub 2020 Nov 5. PMID 33215023
- [Background] Gomez R, Fernandez S, Aspirot A, Punati J, Skaggs B, Mousa H, Di Lorenzo C. Effect of amoxicillin/clavulanate on gastrointestinal motility in children. J Pediatr Gastroenterol Nutr. 2012 Jun;54(6):780-4. doi: 10.1097/MPG.0b013e31824204e4. PMID 22584747
- [Background] Caron F, Ducrotte P, Lerebours E, Colin R, Humbert G, Denis P. Effects of amoxicillin-clavulanate combination on the motility of the small intestine in human beings. Antimicrob Agents Chemother. 1991 Jun;35(6):1085-8. doi: 10.1128/AAC.35.6.1085. PMID 1929247
- [Background] Ciciora SL, Williams KC, Gariepy CE. Effects of Amoxicillin and Clavulanic Acid on the Spontaneous Mechanical Activity of Juvenile Rat Duodenum. J Pediatr Gastroenterol Nutr. 2015 Sep;61(3):340-5. doi: 10.1097/MPG.0000000000000804. PMID 25844706
- [Background] Hulst JM, Zwart H, Hop WC, Joosten KF. Dutch national survey to test the STRONGkids nutritional risk screening tool in hospitalized children. Clin Nutr. 2010 Feb;29(1):106-11. doi: 10.1016/j.clnu.2009.07.006. Epub 2009 Aug 13. PMID 19682776
- [Background] Straney L, Clements A, Parslow RC, Pearson G, Shann F, Alexander J, Slater A; ANZICS Paediatric Study Group and the Paediatric Intensive Care Audit Network. Paediatric index of mortality 3: an updated model for predicting mortality in pediatric intensive care*. Pediatr Crit Care Med. 2013 Sep;14(7):673-81. doi: 10.1097/PCC.0b013e31829760cf. PMID 23863821
- [Derived] Abdelatif RG, Francis AA, Abdelkreem E, Ahmed SH. Amoxicillin for critically ill children with enteral nutrition intolerance (AmoxENI study): A randomized controlled trial. J Pediatr Gastroenterol Nutr. 2025 Sep;81(3):712-721. doi: 10.1002/jpn3.70105. Epub 2025 Jun 12. PMID 40501446